CLINICAL TRIAL: NCT01389284
Title: A Randomized, Double-Blind, Placebo Controlled Trial to Assess the Analgesic Efficacy and Safety of Extended Release Naproxen Sodium Tablets in Postsurgical Dental Pain
Brief Title: Evaluate Efficacy and Safety of Extended Release (ER) Naproxen Sodium
Acronym: VERNE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15142; 2014-005272-28 (EudraCT Number)
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Pain, Postoperative
Keywords: Naproxen Sodium,; dental pain
MeSH Terms: conditions — Pain, Postoperative; Toothache | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Naproxen Sodium ER (BAYH6689) (Experimental): 1 naproxen sodium extended release (ER) 660 mg tablet and 1 naproxen sodium immediate release (IR) 220 mg placebo tablet initially followed by 1 naproxen sodium IR 220 mg matching placebo tablet at hour 8 (± 15 min), and 1 naproxen sodium IR 220 mg matching placebo tablet at hour 16 (± 15 min)
  Interventions: Drug: Naproxen Sodium ER (BAYH6689); Drug: Naproxen Sodium IR Placebo
- Naproxen Sodium IR (Aleve, BAYH6689) (Active Comparator): 1 naproxen sodium ER 660 mg matching placebo tablet and 1 naproxen sodium IR 220 mg tablet initially followed by 1 naproxen sodium IR 220 mg tablet at hour 8 (± 15 min), and 1 naproxen sodium IR 220 mg tablet eight hours at hour 16 (± 15 min)
  Interventions: Drug: Naproxen Sodium IR (Aleve, BAYH6689); Drug: Naproxen Sodium ER Placebo
- Placebo (Placebo Comparator): 1 naproxen sodium ER 660 mg matching placebo tablet and 1 naproxen sodium IR 220 mg matching placebo tablet initially followed by 1 naproxen sodium IR 220 mg matching placebo tablet at hour 8 (± 15 min), and 1 naproxen sodium IR 220 mg matching placebo tablet at hour 16 (± 15 min)
  Interventions: Drug: Naproxen Sodium ER Placebo; Drug: Naproxen Sodium IR Placebo

INTERVENTIONS:
Drug: Naproxen Sodium ER (BAYH6689) — 660 mg Naproxen Sodium extended release tablet, orally administered once daily for 24 hours
  Arms: Naproxen Sodium ER (BAYH6689)
Drug: Naproxen Sodium IR (Aleve, BAYH6689) — 220 mg Naproxen Sodium instant release tablet, orally administered 3 times daily (TID) for 24 hours
  Arms: Naproxen Sodium IR (Aleve, BAYH6689)
Drug: Naproxen Sodium ER Placebo — Matching placebo of 660 mg Naproxen Sodium ER for 24 hours
  Arms: Naproxen Sodium IR (Aleve, BAYH6689); Placebo
Drug: Naproxen Sodium IR Placebo — Matching placebo of 220 mg Naproxen Sodium IR (Aleve) for 24 hours
  Arms: Naproxen Sodium ER (BAYH6689); Placebo

SUMMARY:
The objective is to evaluate pain relief of the extended release naproxen sodium 660 mg tablet compared to commercial naproxen sodium 220 mg tablet over 24 hours in patients with postsurgical dental pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers 15 years of age and above
* Scheduled to undergo surgical removal of up to two impacted third molars, one of which must be mandibular full or partial bony impaction and the other a maxillary impaction
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, NuvaRing, Depo-Provera, or double-barrier and have a negative pregnancy test at Screening and prior to surgery
* Have not taken any form of medication or herbal supplements (ie, St. Johns Wort) within 5 days of admission (except for oral contraceptives, prophylactic antibiotics, or other routine medications to treat benign conditions, such as antibiotics to treat acne) and agree not to take any medication (other than that provided to them) throughout the study
* Have not consumed alcoholic beverages, or foods and beverages containing xanthines (examples, coffee, tea, chocolate, and colas) after midnight prior to surgery and agree not to consume any of these foods or beverages throughout the evaluation period
* Use of only short-acting local anesthetic (e.g., mepivacaine or lidocaine) preoperatively, with or without vasoconstrictor and nitrous oxide
* Have moderate to severe postoperative pain on the Categorical Pain Intensity Scale (a score of at least 2 on a 4 point scale) and a score of ≥ 50 mm on the 100 mm Visual Analog Scale (VAS) within 4 hours postsurgery, but no later than 1330 hours +/- 15 minutes
* Understand the pain rating scales (as judged by the study coordinator)
* Be willing and able to participate in all scheduled visits, treatment plan, tests and other trial procedures according to the protocol
* Provide a personally signed and dated informed consent form (ICF) indicating that the subject has been informed of all pertinent aspects of the trial, (subjects < 18 years of age must sign a written assent and have parental or guardian consent)

Exclusion Criteria:

* History of hypersensitivity to naproxen sodium, acetaminophen, Non Steroidal Anti-inflammatory Drugs (NSAIDS), aspirin, hydrocodone, similar pharmacological agents or components of the investigational products
* Evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, or malignancies within the last 5 years
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted), chronic sinusitis or nasal structural abnormalities causing greater than 50 percent obstruction (polyposis nasi, marked septal deviation) that can interfere with the conduct of the study in the judgment of the investigator
* Current or past history of gastrointestinal bleeding or other bleeding disorder(s)
* Acute illness or local infection prior to surgery that can interfere with the conduct of the study in the judgment of the investigator
* Use of any Over-the-Counter (OTC) or prescription medications with which the administration of naproxen, acetaminophen, ibuprofen or any other NSAIDs, Lortab, is contraindicated or use of any medications within 5 days of surgery (except oral contraceptives, prophylactic antibiotics or medications to treat benign conditions such as antibiotics to treat acne)
* Females who are pregnant or lactating
* Habituation to analgesic drugs (i.e., routine use of oral analgesics 5 or more times per week for greater than 3 weeks)
* Alcoholism or drug abuse within 2 years prior to the Screening Visit or routine consumption of 3 or more alcohol containing beverages per day
* Positive urine, alcohol or nicotine test on day of surgery
* Smokers or using nicotine replacement therapies including transdermal patches, spray, lozenges or gum

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Austin, Texas, United States

REFERENCES:
- [Derived] Laurora I, An R. Efficacy of single-dose, extended-release naproxen sodium 660 mg in postsurgical dental pain: two double-blind, randomized, placebo-controlled trials. Curr Med Res Opin. 2016;32(2):331-42. doi: 10.1185/03007995.2015.1123680. Epub 2015 Dec 15. PMID 26588111
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Started | 120 | 120 | 60
Completed | 120 | 120 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo | Total
Number analyzed (Participants) | 120 | 120 | 60 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.0 (5.05) | 23.0 (4.67) | 25.0 (6.56) | 23.8 (5.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 71 | 41 | 182
  Male | 50 | 49 | 19 | 118
Pain Intensity Score [Number; unit: Participants] — Pain intensity was evaluated using a 4-point Categorical Pain Intensity Rating Scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe
  Participants
    0 = None | 0 | 0 | 0 | 0
    1 = Mild | 0 | 0 | 0 | 0
    2 = Moderate | 96 | 97 | 53 | 246
    3 = Severe | 24 | 23 | 7 | 54

OUTCOME MEASURES:

1. Primary Outcome: Summed, Time-weighted Pain Intensity Difference From 0 to 24 Hours Postdose (SPID0-24)
Description: SPID0-24 was calculated by multiplying the pain intensity difference score at each post-dose timepoint by the duration (in hours) since the preceding timepoint and then summing these values over 0 to 24 hours. Pain intensity was measured at baseline, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 12, 16, 20 and 24 hours using the 4-point categorical pain intensity scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe. SPID0-24 can vary from -24 to 72. The positive SPID value indicates improvement of pain relief. The higher the SPID value, the more improvement of pain relief.
Time Frame: From 0 to 24 hours post-dose
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Error); unit: Score on the scale
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Number analyzed (Participants) | 120 | 120 | 60
Score on the scale | 23.2 (2.01) | 23.6 (2.01) | -0.6 (2.85)

2. Secondary Outcome: Summed, Time-weighted Pain Intensity Differences (SPID)
Description: Pain intensity was measured at baseline, 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 12, 16, 20 and 24 hours using the 4-point categorical pain intensity scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe. The total possible score ranges of SPIDs are SPID0-6: -6 to 18, SPID0-8: -8 to 24, SPID0-12: -12 to 36, SPID0-16: -16 to 48, SPID16-24: -8 to 24. The positive SPID value indicates improvement of pain relief. The higher the SPID value, the more improvement of pain relief.
Time Frame: 0-6, 0-8, 0-12, 0-16 and 16-24 hours postdose
Population: Intent-to-treat (ITT)
Measure: Mean (95% Confidence Interval); unit: Score on the scale
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Number analyzed (Participants) | 120 | 120 | 60
Score on the scale
  From 0 to 6 hours, LS Mean | 5.3 [4.5 to 6.7] | 5.3 [4.5 to 6.1] | -0.5 [-1.6 to 0.7]
  From 0 to 8 hours, LS Mean | 7.0 [5.9 to 8.1] | 6.9 [5.7 to 8.0] | -0.8 [-2.3 to 0.8]
  From 0 to 12 hours, LS Mean | 10.9 [9.1 to 12.7] | 10.9 [9.2 to 12.7] | -0.9 [-3.4 to 1.6]
  From 0 to 16 hours, LS Mean | 14.7 [12.3 to 17.2] | 15.0 [12.5 to 17.5] | -1.0 [-4.5 to 2.6]
  From 16 to 24 hours, LS Mean | 8.5 [6.9 to 10.0] | 8.6 [7.1 to 10.1] | 0.4 [-1.8 to 2.6]

3. Secondary Outcome: Summed, Time-weighted Total Pain Relief Scores (TOTPARs)
Description: TOTPARs were derived by multiplying the pain relief score at each post-dose timepoint by the duration (in hours) since the preceding timepoint and then summing these values over the specified interval. Pain Relief was evaluated at 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 12, 16, 20 and 24 hours postdose, using the 5-point overall pain relief scale: 0 = No relief, 1 = A little relief, 2 = Some relief, 3 = A lot of relief, 4 = Complete relief. The possible total score ranges of TOTPARs are: TOTPAR0-6: 0 to 18, TOTPAR0-8: 0 to 24, TOTPAR0-12: 0 to 36, TOTPAR0-16: 0 to 48, TOTPAR0-24: 0 to 72, TOTPAR16-24: 0 to 24.
Time Frame: 0-6, 0-8, 0-12, 0-16, 0-24, and 16-24 hours postdose
Population: Intent-to-treat (ITT)
Measure: Mean (95% Confidence Interval); unit: Score on the scale
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Number analyzed (Participants) | 120 | 120 | 60
Score on the scale
  From 0 to 6 hours | 13.1 [11.9 to 14.3] | 12.8 [11.6 to 14.0] | 4.7 [2.9 to 6.4]
  From 0 to 8 hours | 17.4 [15.7 to 19.1] | 16.8 [15.1 to 18.5] | 6.1 [3.8 to 8.5]
  From 0 to 12 hours | 26.5 [23.9 to 29.2] | 26.4 [23.7 to 29.0] | 9.7 [5.9 to 13.5]
  From 0 to 16 hours | 35.5 [31.8 to 39.2] | 35.8 [32.0 to 39.5] | 13.4 [8.1 to 18.6]
  From 0 to 24 hours | 54.5 [48.6 to 60.4] | 55.1 [49.2 to 61.0] | 21.8 [13.4 to 30.2]
  From 16 to 24 hours | 19.0 [16.7 to 21.3] | 19.4 [17.1 to 21.6] | 8.4 [5.2 to 11.6]

4. Secondary Outcome: Pain Intensity Differences (PIDs) by Time From Initial Dose
Description: Pain intensity was evaluated using a 4-point Categorical Pain Intensity Rating Scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe
Time Frame: At 0, 0.25, 0.5, 0.75, 1, 2, 3, 4 ,5 ,6, 8, 12, 16, 20 and 24 hours postdose
Population: Intent-to-treat (ITT)
Measure: Mean (95% Confidence Interval); unit: Score on the scale
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Number analyzed (Participants) | 120 | 120 | 60
Score on the scale
  0.25 hours, LS Mean | 1.9 [1.8 to 2.0] | 2.0 [1.9 to 2.1] | 2.0 [1.9 to 2.2]
  0.5 hours, LS Mean | 1.7 [1.6 to 1.8] | 1.7 [1.6 to 1.8] | 1.9 [1.8 to 2.1]
  0.75 hours, LS Mean | 1.4 [1.3 to 1.6] | 1.5 [1.4 to 1.6] | 2.0 [1.8 to 2.2]
  1 hours, LS Mean | 1.2 [1.1 to 1.4] | 1.4 [1.3 to 1.5] | 2.1 [1.9 to 2.3]
  2 hours, LS Mean | 1.2 [1.1 to 1.4] | 1.2 [1.0 to 1.3] | 2.3 [2.1 to 2.5]
  3 hours, LS Mean | 1.2 [1.1 to 1.4] | 1.2 [1.0 to 1.3] | 2.3 [2.1 to 2.6]
  4 hours, LS Mean | 1.2 [1.0 to 1.3] | 1.2 [1.1 to 1.4] | 2.3 [2.1 to 2.5]
  5 hours, LS Mean | 1.3 [1.1 to 1.4] | 1.2 [1.1 to 1.4] | 2.3 [2.1 to 2.5]
  6 hours, LS Mean | 1.3 [1.1 to 1.4] | 1.3 [1.1 to 1.4] | 2.3 [2.1 to 2.5]
  8 hours, LS Mean | 1.3 [1.2 to 1.5] | 1.4 [1.2 to 1.6] | 2.3 [2.1 to 2.6]
  12 hours, LS Mean | 1.2 [1.0 to 1.4] | 1.2 [1.0 to 1.3] | 2.2 [2.0 to 2.5]
  16 hours, LS Mean | 1.2 [1.0 to 1.4] | 1.2 [1.0 to 1.4] | 2.2 [1.9 to 2.5]
  20 hours, LS Mean | 1.2 [1.0 to 1.4] | 1.1 [1.0 to 1.3] | 2.2 [1.9 to 2.5]
  24 hours, LS Mean | 1.1 [0.9 to 1.3] | 1.1 [0.9 to 1.3] | 2.1 [1.8 to 2.3]

5. Secondary Outcome: Pain Relief From Initial Dose
Description: Pain Relief was evaluated using the 5-point overall pain relief scale: 0 = No relief, 1 = A little relief, 2 = Some relief, 3 = A lot of relief, 4 = Complete relief
Time Frame: At 0.25, 0.5, 0.75, 1, 2, 3, 4 ,5 ,6, 8, 12, 16, 20 and 24 hours postdose
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: Score on the scale
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Number analyzed (Participants) | 120 | 120 | 60
Score on the scale
  0.25 hours | 0.9 (0.96) | 0.8 (0.92) | 0.6 (0.75)
  0.5 hours | 1.5 (1.08) | 1.3 (1.02) | 0.8 (0.94)
  0.75 hours | 2.0 (1.21) | 1.7 (1.14) | 0.9 (0.96)
  1 hour | 2.2 (1.29) | 2.0 (1.17) | 0.9 (1.02)
  2 hours | 2.3 (1.30) | 2.3 (1.29) | 0.8 (1.02)
  3 hours | 2.3 (1.33) | 2.4 (1.39) | 0.7 (1.03)
  4 hours | 2.4 (1.41) | 2.2 (1.43) | 0.9 (1.20)
  5 hours | 2.3 (1.35) | 2.2 (1.49) | 0.9 (1.23)
  6 hours | 2.2 (1.37) | 2.2 (1.53) | 0.8 (1.28)
  8 hours | 2.1 (1.40) | 2.0 (1.50) | 0.8 (1.23)
  12 hours | 2.3 (1.51) | 2.4 (1.57) | 0.9 (1.46)
  16 hours | 2.2 (1.52) | 2.3 (1.61) | 1.0 (1.47)
  20 hours | 2.3 (1.58) | 2.3 (1.63) | 1.0 (1.50)
  24 hours | 2.4 (1.63) | 2.5 (1.68) | 1.2 (1.73)

6. Secondary Outcome: Median Time to First Intake of Rescue Medication
Description: Time to first use of rescue medication was estimated using Kaplan-Meier method and analyzed by a logrank test stratified by baseline pain intensity. If at least 50% of subjects in a treatment group took rescue medication, the median time to first rescue was determined for that treatment group.
Time Frame: Up to 24 hours postdose
Population: Intent-to-treat (ITT)
Measure: Median (Full Range); unit: Hours
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Number analyzed (Participants) | 120 | 120 | 60
Hours | NA [NA to NA] — Median Time to Rescue Medication was not computable because less than 50% of the participants did take rescue medication. | NA [NA to NA] — Median Time to Rescue Medication was not computable because less than 50% of the participants did take rescue medication. | 2.9 [1 to 12]

7. Secondary Outcome: Cumulative Percentage of Participants Who Took Rescue Medication
Time Frame: At 0.25, 0.5, 0.75, 1, 2, 3, 4 ,5 ,6, 8, 12, 16, 20 and 24 hours postdose
Population: Intent-to-treat (ITT)
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Number analyzed (Participants) | 120 | 120 | 60
Percentage of participants
  0.25 hours | 0 | 0 | 0
  0.5 hours | 0.0 | 0.0 | 0.0
  0.75 hours | 0.0 | 0.0 | 0.0
  1 hour | 0.0 | 0.0 | 0.0
  2 hours | 7.5 | 7.5 | 30.0
  3 hours | 12.5 | 13.3 | 50.0
  4 hours | 16.7 | 16.7 | 55.0
  5 hours | 18.3 | 20.0 | 58.3
  6 hours | 20.0 | 23.3 | 60.0
  8 hours | 20.8 | 25.0 | 63.3
  12 hours | 22.5 | 25.8 | 66.7
  16 hours | 25.0 | 27.5 | 66.7
  20 hours | 26.7 | 27.5 | 66.7
  24 hours | 26.7 | 27.5 | 66.7

8. Secondary Outcome: Number of Times the Participants Took Rescue Medication Over the 24-hour Period
Time Frame: 24 hours postdose
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: Rescue medication intakes
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Number analyzed (Participants) | 120 | 120 | 60
Rescue medication intakes | 0.5 (0.86) | 0.6 (1.02) | 1.4 (1.20)

9. Secondary Outcome: Global Assessment of the Investigational Product as a Pain Reliever
Description: Global assessment of investigational product as a pain reliever was rated on a 5-point categorical scale: 0 = poor, 1 = fair, 2 = good, 3 = very good, 4 = excellent
Time Frame: 24 hours postdose or immediately before the first intake of rescue medication
Population: Intent-to-treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Number analyzed (Participants) | 120 | 120 | 60
Participants
  0 - Poor | 16 | 18 | 34
  1 - Fair | 14 | 12 | 5
  2 - Good | 22 | 20 | 5
  3 - Very good | 33 | 43 | 12
  4 - Excellent | 35 | 27 | 4

ADVERSE EVENTS:
Arm/Group | Naproxen Sodium ER (BAYH6689) | Naproxen Sodium IR (Aleve, BAYH6689) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120 | 0/60
Other Adverse Events (participants affected / at risk) | 28/120 | 36/120 | 23/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium ER (BAYH6689) (N=120) | Naproxen Sodium IR (Aleve, BAYH6689) (N=120) | Placebo (N=60)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (10) | 9 (9) | 8 (8)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2)
Dental discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tenderness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 6 (6) | 2 (3)
Headache (Nervous system disorders) | 11 (11) | 14 (14) | 12 (12)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 4 (4) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No